CLINICAL TRIAL: NCT00538239
Title: A Pivotal Trial to Determine the Efficacy and Safety of AP23573 When Administered as Maintenance Therapy to Patients With Metastatic Soft-Tissue or Bone Sarcomas
Brief Title: Ridaforolimus in Treatment of Sarcoma-SUCCEED (Sarcoma Multi-Center Clinical Evaluation of the Efficacy of Ridaforolimus)(8669-011 AM6)
Acronym: SUCCEED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8669-011; AP23573-07-302
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Soft-Tissue Sarcomas; Metastatic Bone Sarcomas
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — ridaforolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ridaforolimus (Experimental)
  Interventions: Drug: ridaforolimus
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ridaforolimus — Four 10 mg tablets taken by mouth for 5 days per week continuously
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009
  Arms: Ridaforolimus
Drug: Placebo — Four 10 mg tablets taken by mouth for 5 days per week continuously
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether maintenance therapy with oral AP23573 (ridaforolimus), by preventing and controlling tumor growth for a prolonged period of time in patients with metastatic soft-tissue or bone sarcomas responding to chemotherapy, will result in clinically significant improvement in progression-free survival as compared to oral placebo.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic soft-tissue or bone sarcoma
* Ongoing complete response, partial response, or stable disease (RECIST) after a minimum of 4 cycles (and maximum of 12 months) of any one first, second, or third line of prior cytotoxic chemotherapy for metastatic disease
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate organ and bone marrow function
* Completed prior chemotherapy with last dose received at least 3 and up to 12 weeks prior to randomization

Exclusion Criteria:

* Prior therapy with rapamycin or rapamycin analogs
* Ongoing toxicity associated with prior anticancer therapy
* Another primary malignancy within the past three years
* Concomitant medications that induce or inhibit CYP3A
* Significant, uncontrolled cardiovascular disease

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | Up to 157 weeks after randomization

SECONDARY OUTCOMES:
Overall survival: First Analysis | Up to 157 weeks after randomization
Best Target Lesion Response (RECIST) | Up to 157 weeks after randomization
Overall Survival: Updated Analysis as of 30 April 2011 | Up to 184 weeks after randomization
Overall Survival: Updated Analysis as of 21 January 2012 | Up to 222 weeks after randomization
Safety and tolerability | Up to 157 weeks after randomization

REFERENCES:
- [Result] Demetri GD, Chawla SP, Ray-Coquard I, Le Cesne A, Staddon AP, Milhem MM, Penel N, Riedel RF, Bui-Nguyen B, Cranmer LD, Reichardt P, Bompas E, Alcindor T, Rushing D, Song Y, Lee RM, Ebbinghaus S, Eid JE, Loewy JW, Haluska FG, Dodion PF, Blay JY. Results of an international randomized phase III trial of the mammalian target of rapamycin inhibitor ridaforolimus versus placebo to control metastatic sarcomas in patients after benefit from prior chemotherapy. J Clin Oncol. 2013 Jul 1;31(19):2485-92. doi: 10.1200/JCO.2012.45.5766. Epub 2013 May 28. PMID 23715582